CLINICAL TRIAL: NCT02819258
Title: Monocentric Study and Prognostic of Treatments Endodontics of Teeth With Periapical Pathology Realized CSERD (Nantes University Hospital)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 07/6-N
Record Dates: First submitted 2016-05-31; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Dental Pulp Disorder
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Endodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endodontic treatment for a tooth with a periapical pathology (Other)
  Interventions: Other: Endodontic treatment

INTERVENTIONS:
Other: Endodontic treatment

SUMMARY:
Endodontic therapy is to achieve the eviction of the inflamed or infected pulp and fill the canal opening with a hermetic sealing material.

The analysis of the literature on intracanal therapeutic shows great variability of the results obtained, the reported success rate is 53 to 95%.

This is explained by the difficulty of the surgical procedure, but also by the multiplicity of possible factors of failure, related practitioner, canal anatomy, the operating procedures, the preparation techniques and root canal filling. This success rate is variable depending on the presence or absence of periapical pathology before treatment: more than 85% for teeth treated without initial periapical pathology against only 62% for teeth with pathology before treatment. Furthermore, the literature review revealed two contradictory assumptions about the dominant factor failure in endodontics: the failure of the sealing canal system (bad level shutter) against the failure of the endovascular disinfection.

Main hypothesis of the research objectives:

The probability of success in a year endodontic treatments carried out according to the recommendations and the operating standards on teeth with periapical pathology is approximately 60%.

The primary prognostic factors would be the existence of intracanal obstacles (stop calcification ...) responsible for a sub-obturation of the canal, factors inherent to the tooth (situation ductal anatomy and complexity), the operating techniques used, the practitioner ( skill level), the quality of the restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years
* Patient receiving endodontic treatment for a tooth with a periapical pathology (Category IV of Baume)
* Patients affiliated to a social security scheme or of such a regime,
* Patients admitted to the CSERD,
* Patients in good general health,
* Patient compliant (see medical records: number of appointments not honored)
* Patients with a fixed address and available by telephone, pledging to return a year after treatment at a follow-up consultation for clinical and radiographic examination, and prevent CSERD of any changes of address and telephone number.
* Patients including French
* Patients free of guardianship or trusteeship

Exclusion Criteria:

* Age between 0 and 18
* Tooth with a pulp pathology type Category III of Baume
* Unspecified sheet in diagnosis
* Patients with general contraindication against the endodontic treatment of teeth with periapical pathology (risk oslérien, immuno-depressed subjects, patients with prosthetic hip, knee).
* No possibility of rubber dam during endodontic treatment.
* Patient with latex allergy (contraindicating the installation of a dam and possibly endodontic obturation with gutta-percha)
* Patients whose postoperative follow is deemed random by the investigator (cf. medical record: number of appointments not honored)
* Patient not engaging to return for clinical and radiographic examination in a year
* Patients with temporary housing or no fixed address: Living in a furnished accommodation or a hotel room, in a nursing home, in a home-type squat, Homeless
* Patients not meeting all inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The assessment at one year of intracanal treatment on teeth defined on clinical and radiographic criteria, as recommended by the ESE (European Society of Endodontology) (success / failure / uncertain cases) | 1 year
  Consider the probability of failure of intracanal treatment on teeth with periapical pathology in the first year following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Benedicte ENKEL, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France